

## SYNFIX. A cohort study of Bioabsorbable screws for Syndesmosis Fixation in Ankle Fractures

Chief Investigator: Professor Alan Johnstone

IRAS project number 209339. REC Ref: 17/NS/0068

Copies: 1 for Patient; 1 for Researcher; 1 to be filed within Patient's Hospital Notes

| INFORMED CONSENT FORM | | Participant ID | |
|---|---|---|---|
| | | P | lease initial box |
| 1. I confirm that I have read and u | nderstand the infor | mation sheet Version dated// | |
| for the above clinical trial and have | e had the opportun | ity to consider the information, ask | |
| questions and have had these ans | wered satisfactorily | <i>'</i> . | |
| 2. I understand that my participat | ion in this clinical tr | ial is voluntary and that I am free to withdraw | <i>,</i> |
| at any time and without giving an | y reason, without m | ny medical care or legal rights being affected. | |
| Data collected up until the point of | withdrawal may still | I be used in analysis. | |
| the clinical study may be looked a | t by responsible ind<br>t to my taking part i | y medical notes and data collected during<br>lividuals from regulatory authorities or from<br>n this research. I give permission for these | |
| 4. I agree for my information to be | stored on NHS Gra | mpian servers. | |
| 5. I agree to participate in the above study. | | | |
| Name of Patient | Date | Signature | |
| Name of Person taking consent | Date | Signature | |
| Researcher | <br>Date | Signature | |